CLINICAL TRIAL: NCT05036499
Title: Development of a Personalized Feedback Intervention Targeting Pain-Related Anxiety for Hazardous Drinkers With Chronic Pain
Brief Title: PFI for Pain-Related Anxiety Among Hazardous Drinkers With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Andrew Rogers, Principal Investigator, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F31AA028694 (NIH); F31AA028694 (NIH)
Record Dates: First submitted 2021-08-06; First posted 2021-09-05 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Alcohol Problem; Chronic Pain; Alcohol Abuse
MeSH Terms: conditions — Alcohol-Related Disorders; Chronic Pain; Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Feedback Intervention (PFI) (Experimental): Personalized Feedback Intervention targeting pain-related anxiety for hazardous drinkers with chronic pain
  Interventions: Behavioral: Personalized Feedback Intervention
- Assessment Only (No Intervention): Assessment only, no active treatment elements

INTERVENTIONS:
Behavioral: Personalized Feedback Intervention — Providing corrective normative feedback on alcohol use, psychoeducation on the interplay between pain and alcohol use, and providing exercises to target pain-related anxiety
  Arms: Personalized Feedback Intervention (PFI)

SUMMARY:
There is a pressing public health need to develop novel interventions that aim to reduce alcohol consumption and concurrent alcohol among hazardous drinkers with comorbid chronic pain. The proposed study will draw upon NIH treatment development guidelines (Stage 1) to translate and innovate past work to address a major public health priority. Specifically, we propose to develop (Phase IA) and pilot test (Phase IB) a brief, integrated, single-session, computer-based personalized feedback intervention (PFI) designed to 1) enhance knowledge regarding adverse pain-related anxiety-alcohol interrelations; and (2) increase motivation and intention to reduce hazardous drinking.

DETAILED DESCRIPTION:
Hazardous alcohol use contributes to mental and physical health problems, disability, and may lead to increased risk of premature death. Among individuals with chronic pain the rate of hazardous alcohol use is elevated compared to the general population, yet, hazardous alcohol users with chronic pain remain an underserved group. There is a critical need to test alternative and complimentary approaches to the implementation of effective interventions to reduce hazardous alcohol use among this high-risk segment of the general population; doing so in an integrated fashion (i.e., jointly targeting alcohol and affective mechanisms that may maintain pain-alcohol associations) may provide a more efficient and targeted intervention approach. Targeting pain-related anxiety, a transdiagnostic vulnerability factor that is prospectively associated with both hazardous drinking and chronic pain, may be beneficial. Thus, more work is needed to evaluate the benefit of targeting elevated pain-related anxiety among hazardous drinkers with chronic pain. Our approach will follow a staged model consistent with NIH guidelines for developing and standardizing behavioral interventions. Phase IB activities will include a proof-of-concept and highly rigorous randomized clinical trial designed to compare pain-related anxiety/alcohol PFI (PA-PFI) to assessment only among a sample of 130 hazardous drinkers with chronic pain who have elevated levels of pain-related anxiety. This study represents an important and pivotal step in the larger landscape of translating basic research to more efficacious strategies for reducing hazardous drinking among underserved populations with medical comorbidities. The proposed intervention would be highly disseminable and relevant to millions of hazardous drinkers with chronic pain. Given the collective public health impact of chronic pain and hazardous drinking, the proposed study will yield findings that enhance scientific knowledge, enhance our understanding of mechanisms in reciprocal pain-alcohol relations, and inform the development of novel treatments for hazardous drinkers with chronic pain with elevated pain-related anxiety that are adaptable and easily implemented across a variety of healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 21 years of age
* Current hazardous drinking pattern (AUDIT scores ≥ 8 for males and ≥ 7 for females)
* Current chronic pain (1) on most days of the week (i.e., 4 or more days per week), (2) at an average weekly severity of 3 or greater on a 0-10 numerical rating scale, and (3) for at least three months in duration
* Fluent in English

Exclusion Criteria:

1. Concurrent alcohol or other substance use treatment
2. Not being fluent in English
3. Current acute psychiatric distress or thought disorder
4. Current imminent risk of suicidality

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Hazardous Drinking | 2 weeks post intervention
  Alcohol Use Disorders Identification Test - Scores below 8 (males) and 7 (females) indicate non-hazardous drinking
Hazardous Drinking | 1 month post intervention
  Alcohol Use Disorders Identification Test - Scores below 8 (males) and 7 (females) indicate non-hazardous drinking
Drinking Quantitiy/Frequency | 2 weeks post intervention
  Timeline Follow Back will be used to assess past 2 week drinking quantity and frequency, and an average alcohol consumption variable will be created
Drinking Quantitiy/Frequency | 1 month post intervention
  Timeline Follow Back will be used to assess past 2 week drinking quantity and frequency, and an average alcohol consumption variable will be created

SECONDARY OUTCOMES:
Pain-related Anxiety | Immediately Post intervention
  A measure of anxiety related to pain (pain anxiety symptoms scale 20) and pain-elicitnig activities. Range of scores from 0-100, with higher scores indicating greater fear and anxiety.
Pain-related Anxiety | 2 weeks post intervention
  A measure of anxiety related to pain (pain anxiety symptoms scale 20) and pain-elicitnig activities. Range of scores from 0-100, with higher scores indicating greater fear and anxiety.
Pain-related Anxiety | 1 month post intervention
  A measure of anxiety related to pain (pain anxiety symptoms scale 20) and pain-elicitnig activities. Range of scores from 0-100, with higher scores indicating greater fear and anxiety.
Motivation to Reduce Drinking | Immediately Post intervention
  The Alcohol Ladder will be used to assess motivation to reduce drinking on a 0-10 scale, with 0 indicating no motivation to reduce drinking, and 10 indicating 100% intend to reduce drinking.
Motivation to Reduce Drinking | 2 weeks post intervention
  The Alcohol Ladder will be used to assess motivation to reduce drinking on a 0-10 scale, with 0 indicating no motivation to reduce drinking, and 10 indicating 100% intend to reduce drinking.
Motivation to Reduce Drinking | 1 month post intervention
  The Alcohol Ladder will be used to assess motivation to reduce drinking on a 0-10 scale, with 0 indicating no motivation to reduce drinking, and 10 indicating 100% intend to reduce drinking.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Zvolensky, Ph.D., Study Chair — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No